CLINICAL TRIAL: NCT02971059
Title: Phenylalanine Requirement of Healthy Older Adult Males and Females > 65 Years Determined by Direct Amino Acid Oxidation (DAAO) Method.
Brief Title: Phenylalanine Requirement of Adults >65 Years.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Project Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1000051682
Record Dates: First submitted 2016-11-14; First posted 2016-11-22 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Older Adults
Keywords: Elderly; Phenylalanine; Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adult Males >65 years (Experimental): Participants will be seen initially for pre-study assessment (3 hour). They will then be studied weekly for up to 7 levels of phenylalanine intake (7 Study periods). Each study period will include a period of 3 days. The first 2 days they will consume a liquid milkshake based diet at home. On the 3rd day they will come to the hospital for a total of 8 hours.
  Interventions: Dietary Supplement: Phenylalanine intake
- Adult Females >65 years (Experimental): Participants will be seen initially for pre-study assessment (3 hour). They will then be studied weekly for up to 7 levels of phenylalanine intake (7 Study periods). Each study period will include a period of 3 days. The first 2 days they will consume a liquid milkshake based diet at home. On the 3rd day they will come to the hospital for a total of 8 hours.
  Interventions: Dietary Supplement: Phenylalanine intake

INTERVENTIONS:
Dietary Supplement: Phenylalanine intake — Phenylalanine will be provided as graded intakes ranging from 7-40 mg/kg/day

SUMMARY:
Currently there are insufficient published studies on amino acid requirements in the elderly. Phenylalanine is one of the indispensable amino acids. Low levels of phenylalanine has been observed in in the blood of older adults. It is due the increased uptake by the liver and intestine. This decreased levels of phenylalanine could lead to decreased skeletal muscle protein synthesis. Requirement for elderly individuals have been set based on studies conducted in younger adults hence may be inaccurate. The goal of this study is to directly measure the phenylalanine requirement of male and female elderly subjects over 65 years using the direct amino acid oxidation (DAAO) technique.

DETAILED DESCRIPTION:
1. To determine and compare the phenylalanine requirement of healthy elderly male and female adults over the age of 65 years using the DAAO technique (by measuring the oxidation of L-[1-13 C] phenylalanine to 13 CO 2 [F 13 CO 2] ) in response to graded intakes of phenylalanine.
2. To compare the requirement so derived to that of young healthy adult previously determined in our lab.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy elderly males and females > 65 years
2. Willingness to participate in the study and completed the screening procedures (height, weight, fasting blood sample and medical history questionnaire).
3. No recent history of weight loss
4. Absence of chronic disease or acute illness that could affect protein and AA metabolism (diabetes, cancer, liver or kidney disease, HIV, acute cold or flu, hypo or hyperthyroidism, rheumatoid arthritis treated with anti-inflammatory medications.
5. Non-smoking
6. Willingness to consume the diet provided

Exclusion Criteria:

1. Presence of disease known to affect protein and AA metabolism (diabetes, cancer, liver or kidney disease, HIV, acute cold or flu, hypo or hyperthyroidism, rheumatoid arthritis treated with anti-inflammatory medications).
2. On medications known to affect protein and amino acid metabolism (steroids).
3. Recent significant weight loss.
4. Individual on weight reducing diets.
5. Inability to tolerate the diet
6. Unwilling to have blood drawn from a venous access, or using a ventilated hood indirect calorimeter for the purposes of the study.
7. Significant coffee consumption of more than 2 cups/day
8. Significant alcohol consumption of more than one drink/day

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Phenylalanine Requirement | Baseline
  To determine phenylalanine requirement by measuring the oxidation of 13CO2 in breath in response to graded phenylalanine intakes

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, Principal Investigator — Hospital for Sick Children, Toronto, Ontario
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin KE, Pencharz PB, Rafii M, Ball RO, Szwiega S, Elango R, Courtney-Martin G. The Phenylalanine Requirement of Elderly Men and Women Measured by Direct 13C Carbon Oxidation Method Is Similar to That of Young Adults. J Nutr. 2019 Oct 1;149(10):1776-1784. doi: 10.1093/jn/nxz137. PMID 31271193